CLINICAL TRIAL: NCT04743882
Title: A Comparison of the Analysis of the Force on the Supporting Legs of Female Athletes of Different Levels Playing Football
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, yecheng zhang, Biomechanics Laboratory, Universidad Politecnica de Madrid
Other Study IDs: UPMadrid-Yecheng.Zhang
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Condition Angle, Angular Velocity, Linear Velocity, Moment, Ground Reaction Force, Hip Joint, Knee Joint, Ankle Joint

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A
- B
- C

INTERVENTIONS:
Other:

SUMMARY:
In this study, we grouped athletes into different training levels, and tested the force on the supporting legs of female athletes at different times when they kicked the ball.

DETAILED DESCRIPTION:
In this study, first we divided the subjects into three levels: A, B, and C. After fully warming up, we asked the subjects to perform five full kicks. The kicking process was captured with a Vicon high-speed camera. The data captured by the motion capture system was then analyzed to analyze the angles, angular velocity, linear velocity, and ground reaction force of the hip, knee, and ankle joints of the hip, knee, and ankle supporting legs of female athletes of different levels during full kicks. Finally, the subjects of different levels are analyzed to find the significant differences in the supporting legs of female football players of different levels.

ELIGIBILITY:
Inclusion Criteria:

* Master kicking skills Have not suffered any injury of lower limbs in the past six months

Exclusion Criteria:

* Unable to complete the kick Has suffered a lower limb injury in the past six months

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female athletes with good kicking skills
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
hip | 1month
  Analysis of hip angle and angular velocity of ABC three groups of athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- UPM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Analyze the force on the lower limbs of female football players of different levels